CLINICAL TRIAL: NCT02234531
Title: Assessment of a Virtual Teacher Feedback for the Recovery of Upper Limb After Stroke.
Brief Title: Comparison Study of 'Virtual Teacher' Support for Rehabilitation After Stroke.
Acronym: MAVASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: Società Italiana di Fisioterapia (SIF) (Unknown); Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Andrea Turolla, PhD, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocollo 2013.11
Record Dates: First submitted 2014-08-29; First posted 2014-09-09 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: Virtual Reality,; Enhanced Feedback,; Stroke,; Rehabilitation,; Motor Learning
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVER TEACHER (Experimental): In EVER TEACHER group a specific feedback called "virtual teacher" will be displayed. The virtual teacher perform the correct movement to emulate, that is supposed to stimulate the motor adaptation exploiting a supervised learning mechanism. This feedback will give an on-line information on motor performance quality, allowing a real time visual comparison between patient's own execution and teacher one. During the experiment, patients will receive 1 hour of virtual reality-based therapy and the treatment will last 1 hour a day, five days weekly for four weeks.
  Interventions: Device: EVER TEACHER
- NEVER TEACHER (Other): In NEVER TEACHER group the subjects will be asked to perform the same exercises with the upper limb without the virtual teacher assistance. The treatment will last four weeks with daily sessions of 60 minutes, five times per week.
  Interventions: Device: NEVER TEACHER

INTERVENTIONS:
Device: EVER TEACHER — The treatment will be performed in a darkened room, to avoid distraction provided by environmental stimuli. The patients will be seat on a standard chair in front of a wall screen handling a sensorized object with plegic hand. In case of grasping deficits the hand's surface will be used as end effector (i.e. sensorized glove worn by the patient). During the treatment a specific feedback called "virtual teacher" will be displayed. The Reinforced Feedback in Virtual Environment (RFVE) approach consists of performing different motor tasks moving the end effector simultaneously displayed in the virtual scenario. The Virtual Reality Rehabilitation System (VRRS®. Khymeia Group, Noventa Padovana. Italy) will be used as device to provide the artificial environment.
  Arms: EVER TEACHER
Device: NEVER TEACHER — The patients allocated to NEVER TEACHER group, will be treated using the VRRS and the proceedings will be the same as described for experimental group. In this group, the patient will move the real object (e.g. ball) following the trajectory of the corresponding virtual object displayed on the wall screen in accordance with the requested virtual task and without the 'virtual teacher' support.
  Arms: NEVER TEACHER

SUMMARY:
The aim of the project is to assess whether the continuous visualization of on-line teacher in virtual reality (VR) is effective for the improvement of upper limb motor function, in stroke patients.

DETAILED DESCRIPTION:
A single-blind randomized controlled trial (RCT) will be carried out to compare the effects of reinforced feedback in virtual environment (RFVE) treatment with continuous displaying of a virtual teacher (EVER TEACHER group) with RFVE without the presence of a virtual teacher (NEVER TEACHER group).

ELIGIBILITY:
Inclusion Criteria:

* first single stroke,
* absence of ideomotor apraxia, neglect, aphasia interfering with verbal comprehension,
* 0 < NIHSS-IT < 4

Exclusion Criteria:

* bilateral or cerebellum stroke,
* unstable medical conditions,
* fracture,
* major depressive disorders,
* other neurological conditions,
* epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity scale (FM UE) | Change from baseline FM UE scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - Sensation | Change from baseline of the Reaching Performance scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).
Fugl-Meyer Assessment - Pain and ROM | Change from baseline of the Reaching Performance scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).
Reaching Performance Scale | Change from baseline of the Reaching Performance scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).
Modified Ashworth Scale | Change from baseline of the Modified Ashworth scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).
Functional Independence Measure scale (FIM) | Change from baseline of the Functional Independence Measure scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).
Nine Hole Pegboard Test | Change from baseline of the Functional Independence Measure scale at the end of Virtual therapy (four weeks thereafter)
  Applied at the beginning and at the end of treatment (after 20 sessions).

OTHER OUTCOMES:
Kinematic Assessment | Change from baseline of the following parameters; speed, time, peak at the end of Virtual therapy (four weeks thereafter)
  The kinematic assessment include the execution of standardised upper limb movements, such as: forearm pronation and supination, elbow flexion and extension, shoulder abduction and adduction, shoulder internal and external rotation, shoulder flexion and extension and reaching movements. The mean linear velocity (Speed), the mean duration of movements (Time) and the mean number of submovements (Peak) will be measured, by means of the Virtual Reality Rehabilitation System (VRRS®. Khymeia Group, Noventa Padovana. Italy). The data will be registered at the beginning and at the end of treatment, 4 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — San Camillo IRCCS
Locations (2):
- Italy (2):
  - San Camillo IRCCS, Venezia, VE
  - Azienda ULSS 3 Serenissima, Venice

REFERENCES:
- [Background] Turolla A, Dam M, Ventura L, Tonin P, Agostini M, Zucconi C, Kiper P, Cagnin A, Piron L. Virtual reality for the rehabilitation of the upper limb motor function after stroke: a prospective controlled trial. J Neuroeng Rehabil. 2013 Aug 1;10:85. doi: 10.1186/1743-0003-10-85. PMID 23914733
- [Background] Kiper P, Agostini M, Luque-Moreno C, Tonin P, Turolla A. Reinforced feedback in virtual environment for rehabilitation of upper extremity dysfunction after stroke: preliminary data from a randomized controlled trial. Biomed Res Int. 2014;2014:752128. doi: 10.1155/2014/752128. Epub 2014 Mar 13. PMID 24745024
- [Background] Zucconi C, Valt V, Agostini M, Turolla A, Tonin P, Piron L. Assessment of a virtual teacher feedback for the recovery of the upper limb after stroke. Italian Journal of Physiotherapy 2011;1(4):101-6.
- See also: Italian Society for Physiotherapy (Società Italiana di Fisioterapia) — http://www.sif-fisioterapia.it/